CLINICAL TRIAL: NCT01449630
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety and Tolerability of LY3031207 in Healthy Subjects
Brief Title: A Study of LY3031207 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14283; I5W-EW-LBCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY3031207; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3031207 (Experimental): Participants received escalating doses of 5 mg (milligrams), 25 mg, 75 mg, 225 mg, 450 mg and 900 mg of LY3031207 capsule orally.
  Interventions: Drug: LY3031207
- Placebo (Placebo Comparator): Single dose of placebo administered orally in up to two occasions separated by at least a 3 week wash-out period between each dose.
  Interventions: Drug: Placebo
- Celecoxib (Active Comparator): Single 400mg dose of celecoxib administered orally on one occasion.
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: LY3031207 — Administered orally
  Arms: LY3031207
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Celecoxib — Administered orally
  Arms: Celecoxib

SUMMARY:
This is a phase I study of LY3031207 in healthy subjects. The purposes of this study are to look at safety, how well the study drug is tolerated, and how much of the study drug gets into the blood stream and how long it takes the body to get rid of it when given to humans. Information about any side effects that may occur will also be collected. Subjects will participate in the study for approximately 3 months. This study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects agree to use a reliable method of birth control during the study and for 3 months following the last dose of the investigational product
* Women not of child-bearing potential due to surgical sterilization (at least 6 weeks after surgical bilateral oophorectomy with or without hysterectomy or at least 6 weeks after tubal ligation) confirmed by medical history or menopause
* Menopausal women include women with either spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications during the amenorrhea that induced the amenorrhea (for example [e.g.], oral contraceptives, hormones, gonadotropin-releasing hormone, antiestrogens, selective estrogen receptor modulators, or chemotherapy) or spontaneous amenorrhea for 6 to 12 months and a follicle-stimulating hormone level greater than 40 milli-International Unit (mIU/mL)
* Overtly healthy based on the history and physical examinations as determined by the investigator
* Between body mass index (BMI) of 18.5 and 32.0 kilogram per meter squared (kg/m^2), inclusive
* Normotensive defined as supine systolic blood pressure (BP) <140 of millimeter mercury (mmHg), and diastolic BP <90 mmHg, without the use of any antihypertensives, or results that are judged to be not clinically significant by the Investigator. Blood pressure may be retested up to 2 additional times, under well rested conditions
* Clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Ex vivo whole blood prostaglandin E(PGE) synthesis after lipopolysaccharide (LPS) stimulation of no less than 5 nanograms/milliliter (ng/mL).
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product or unapproved use of a drug with a short half-life, or within 5 half-life of an investigational product with a half-life longer than 5 days, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have known allergies to LY3031207 or any components of the formulation, celecoxib or sulfonamides. Subjects with known aspirin allergy or allergic reaction to non-steroidal anti-inflammatory drugs (NSAIDs) should also be excluded
* Are persons who have previously completed or withdrawn from this study or any other study investigating LY3031207 and who have previously received the investigational product
* Have an abnormality in the 12-lead Electrocardiogram (ECG), including QTc interval with Bazett's correction >450 millisecond (msec) for men and >470 msec for women or an abnormality that, in the opinion of the investigator, increases the risks associated with participating in the study. Electrocardiogram may be repeated after 5 minutes resting quietly, if the subject's heart rate is >75 beats per minute
* History of, within the last 2 years, or presence of active cardiovascular disease, including acute myocardial infarction, unstable angina, congestive heart failure, stroke, or transient ischemic attack
* Presence of clinically significant active bleeding or history of bleeding diathesis at the time of screening
* Presence of active peptic ulcer disease, Gastrointestinal (GI) bleeding, chronic gastritis, inflammatory bowel disease, chronic diarrhea, or positive H. pylori serology
* Evidence of hepatitis C and/or positive hepatitis C antibody
* Evidence of hepatitis B and/or positive hepatitis B surface antigen
* Evidence of other chronic liver disease, including chronic alcoholic disease; non-alcoholic steatohepatitis; recent (within 3 months of screening) history of acute viral hepatitis; or subjects with known Gilbert Syndrome
* History of active neuropsychiatric disease
* Evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* Have a significant history of or current other cardiovascular, respiratory (especially asthma and chronic obstructive pulmonary disease), hepatic, renal, GI, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data. History of prior surgeries (at least 3 months prior to dosing), such as splenectomy, cholecystectomy, and appendectomy are not exclusionary
* Regularly use of known drugs of abuse and/or show positive findings on urinary drug screening
* Are women with a positive pregnancy test or women who are lactating
* Intended use of over-the-counter medications or prescription medication within 14 days prior to dosing, this includes but is not limited to antihypertensives, diuretics, antiplatelet or anticoagulant drugs, and antidepressants
* Any use of NSAIDs, celecoxib, aspirin or acetaminophen (at doses >1 gram [gm] per day) within 14 days of screening
* Any use of herbal or dietary supplements, or grapefruit and/or grapefruit juice, Seville oranges, starfruit, or pomegranate within 14 days prior to dosing of study drug
* Have donated blood of more than 500 milliliter (mL) within the last month
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 ounce [oz] or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Subjects who smoke more than 10 cigarettes per day or are unwilling to follow the Clinical Research Unit (CRU) smoking rules
* Subjects with any major surgery within 30 days prior to screening or subjects with planned surgeries to occur during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-10-24 (Actual); Primary Completion 2012-04-02 (Actual); Study Completion 2012-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three period crossover study with three dosing cohorts. The interval between the initiation of each dosing cohort was approximately 1 week, and the washout time between each dosing period was approximately 3 weeks.
Groups:
- Cohort I Sequence 1: Participants received 5 mg LY3031207, Placebo and 400 mg Celecoxib as per the below dosing schedule.
  Period 1: 5 mg LY3031207 , Period 2: Placebo, and Period 3: 400 mg Celecoxib
- Cohort I Sequence 2: Participants received 5 mg LY3031207, 225 mg LY3031207 and 400 mg Celecoxib as per the below dosing schedule.
  Period 1: 5 mg LY3031207, Period 2: 225 mg LY3031207 and Period 3: 400 mg Celecoxib
- Cohort I Sequence 3: Participants received Placebo, 225 mg LY3031207 and 400 mg Celecoxib as per the below dosing schedule.
  Period 1: Placebo, Period 2: 225 mg LY3031207 and Period 3: 400 mg Celecoxib
- Cohort II Sequence 1: Participants received 25 mg LY3031207 and Placebo as per the below dosing schedule.
  Period 1: 25 mg LY3031207, Period 2: Placebo and Period 3: Placebo
- Cohort II Sequence 2: Participants received 25 mg LY3031207, 450 mg LY3031207 (Fed condition) and 450 mg LY3031207 (Fasted) as per the below dosing schedule.
  Period 1: 25 mg LY3031207, Period 2: 450 mg LY3031207 (Fed) and Period 3: 450 mg LY3031207 (Fasted)
- Cohort II Sequence 3: Participants received Placebo, 450 mg LY3031207 (Fed condition) and 450 mg LY3031207 (Fasted) as per the below dosing schedule.
  Period 1: Placebo, Period 2: 450 mg LY3031207 (Fed) and Period 3: 450 mg LY3031207 (Fasted)
- Cohort III Sequence 1: Participants received LY3031207 75 mg, Placebo and celecoxib as per the below dosing schedule.
  Period 1: LY3031207 75 mg, Period 2: Placebo and Period 3: Celecoxib 400 mg
- Cohort III Sequence 2: Participants received LY3031207 75 mg, LY3031207 900 mg and celecoxib as per the below dosing schedule.
  Period 1: LY3031207 75 mg, Period 2: LY3031207 900 mg and Period 3: Celecoxib 400 mg
- Cohort III Sequence 3: Participants received Placebo, LY3031207 900 mg and celecoxib as per the below dosing schedule.
  Period 1: Placebo, Period 2: LY3031207 900 mg and Period 3: Celecoxib 400 mg
Period: Period 1
Arm/Group | Cohort I Sequence 1 | Cohort I Sequence 2 | Cohort I Sequence 3 | Cohort II Sequence 1 | Cohort II Sequence 2 | Cohort II Sequence 3 | Cohort III Sequence 1 | Cohort III Sequence 2 | Cohort III Sequence 3
Started | 2 | 6 | 2 | 2 | 5 | 2 | 2 | 6 | 2
Received at Least 1 Dose | 2 | 6 | 2 | 2 | 5 | 1 | 2 | 6 | 2
Completed | 1 | 6 | 2 | 1 | 5 | 1 | 2 | 6 | 2
Not Completed | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort I Sequence 1 | Cohort I Sequence 2 | Cohort I Sequence 3 | Cohort II Sequence 1 | Cohort II Sequence 2 | Cohort II Sequence 3 | Cohort III Sequence 1 | Cohort III Sequence 2 | Cohort III Sequence 3
Started | 1 | 6 | 2 | 1 | 5 | 1 | 2 | 6 | 2
Completed | 1 | 6 | 2 | 1 | 5 | 1 | 1 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Cohort I Sequence 1 | Cohort I Sequence 2 | Cohort I Sequence 3 | Cohort II Sequence 1 | Cohort II Sequence 2 | Cohort II Sequence 3 | Cohort III Sequence 1 | Cohort III Sequence 2 | Cohort III Sequence 3
Started | 1 | 6 | 2 | 1 | 5 | 1 | 1 | 6 | 2
Completed | 1 | 6 | 2 | 1 | 5 | 1 | 1 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I Sequence 1 | Cohort I Sequence 2 | Cohort I Sequence 3 | Cohort II Sequence 1 | Cohort II Sequence 2 | Cohort II Sequence 3 | Cohort III Sequence 1 | Cohort III Sequence 2 | Cohort III Sequence 3 | Total
Number analyzed (Participants) | 2 | 6 | 2 | 2 | 5 | 2 | 2 | 6 | 2 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 2 | 2 | 5 | 2 | 2 | 6 | 2 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 9
  Male | 1 | 3 | 1 | 2 | 4 | 1 | 1 | 5 | 2 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  White | 1 | 6 | 2 | 2 | 4 | 2 | 2 | 6 | 1 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 6 | 2 | 2 | 5 | 2 | 2 | 6 | 2 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Drug Related Adverse Events (AE) or Any Serious AE
Description: AEs that were considered possibly related to study drug, in the opinion of the investigator, were reported. A summary of serious and all other non-serious AEs, regardless of possible drug relatedness, is located in the Reported Adverse Event module.
Time Frame: Baseline, up to 4 months
Population: All participants who received at least 1 dose of study drug or placebo.
Measure: Count of Participants; unit: Participants
Groups:
- 5 mg LY3031207: 5 milligrams (mg) LY3031207 administered orally as capsules as a single dose.
- 25 mg LY3031207: 25 mg LY3031207 administered orally as capsules as a single dose.
- 75 mg LY3031207: 75 mg LY3031207 administered orally as capsules as a single dose.
- 225 mg LY3031207: 225 mg LY3031207 administered orally as capsules as a single dose.
- 450 mg LY3031207 Fed: 450 mg LY3031207 administered orally as capsules as a single dose.
- 450 mg LY3031207 Fasted: 450 mg LY3031207 administered orally as capsules as a single dose to participants who were fasted.
- 900 mg LY3031207: 900 mg LY3031207 administered orally as capsules as a single dose.
- Placebo: Matched placebo capsules administered orally.
- 400 mg Celecoxib: 400 mg Celecoxib administered orally as capsules.
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207 | Placebo | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8 | 10 | 18
Participants
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other Non-Serious AEs | 3 | 3 | 1 | 1 | 0 | 2 | 2 | 2 | 1

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of LY3031207
Description: AUC from time 0 to last timepoint (AUC0-tlast) with measurable concentration of LY3031207.
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 96, 144 hours post dose
Population: Pharmacokinetic (PK) population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- 5 mg LY3031207: 5 mg LY3031207 administered orally as capsules as a single dose.
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8
nanogram*hour per milliliter (ng*hr/mL) | 3040 (31) | 13900 (65) | 40000 (32) | 151000 (28) | 171000 (54) | 116000 (73) | 348000 (63)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3031207
Time Frame: Predose, 0.25, 0.5, 1, 2, 4, 8, 12, 24, 48, 96, 144 hours post dose
Population: Pharmacokinetic (PK) population: all participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8
nanograms per milliliter (ng/mL) | 185 (35) | 818 (40) | 2060 (20) | 5610 (31) | 7780 (32) | 5670 (49) | 11300 (45)

4. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Ex Vivo Whole Blood Prostaglandin E (PGE) Synthesis After Lipopolysaccharide (LPS) Stimulation
Description: The effect of LY3031207 on PGE synthesis in whole blood after ex vivo LPS stimulation.
Time Frame: Predose, 0.5, 1, 2, 8, 24 and 144 hours post dose.
Population: All participants who received at least 1 dose of study drug or placebo with evaluable PGE data at the specific time points.
Measure: Mean (Standard Deviation); unit: percentage change in PGE
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207 | Placebo | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 18
percentage change in PGE
  0.5 hours (hr): number analyzed (Participants) | 8 | 5 | 8 | 7 | 5 | 6 | 8 | 11 | 18
  0.5 hours (hr) | -16.2 (32.9) | -15.6 (26.4) | 33.0 (45.0) | 12.7 (64.0) | 42.7 (69.7) | -85.1 (13.8) | -43.1 (17.8) | 56.1 (97.9) | -10.4 (77.6)
  1 hr: number analyzed (Participants) | 7 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 17
  1 hr | -9.2 (43.5) | -4.8 (67.7) | 24.6 (67.5) | -16.8 (93.7) | -83.8 (41.4) | -92.9 (8.5) | -93.7 (6.9) | 65.4 (116.8) | -44.8 (59.5)
  2 hr: number analyzed (Participants) | 7 | 6 | 8 | 6 | 6 | 6 | 8 | 10 | 18
  2 hr | -34.3 (20.1) | -45.5 (49.4) | -47.0 (19.8) | -79.2 (21.2) | -104.9 (11.8) | -96.4 (8.9) | -83.3 (11.8) | 65.1 (106.6) | -68.2 (27.8)
  8 hr: number analyzed (Participants) | 8 | 6 | 8 | 6 | 6 | 6 | 6 | 11 | 15
  8 hr | -8.5 (41.0) | -40.1 (25.4) | -41.3 (35.9) | -79.3 (6.6) | -94.3 (13.9) | -88.3 (13.5) | -98.4 (3.8) | 76.9 (109.1) | -63.1 (32.1)
  24 hr: number analyzed (Participants) | 8 | 6 | 8 | 1 | 6 | 6 | 8 | 9 | 18
  24 hr | 89.4 (153.9) | 8.7 (73.3) | 60.0 (84.3) | -29.5 (NA) — Not analyzed due to insufficient number of participants. | -76.8 (40.6) | -54.1 (28.4) | -88.8 (12.2) | 124.8 (139.3) | -19.9 (60.7)
  144 hr: number analyzed (Participants) | 7 | 6 | 7 | 7 | 3 | 6 | 8 | 11 | 16
  144 hr | 178.2 (96.5) | 24.3 (58.2) | 153.7 (70.9) | 131.1 (111.4) | 125.1 (104.6) | 48.0 (49.3) | 41.4 (101.1) | 159.1 (138.7) | 7.6 (76.5)

5. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Urinary Excretion of Prostaglandin E(2) Metabolite (PGEM)
Description: The participant's urine was collected during protocol-defined intervals and the PGE metabolite PGEM was assessed. PGEM results for each interval were then compared to the baseline value.
Time Frame: 0 to 2, 2 to 4, 4 to 6, 6 to 12 and 12 to 24 hours post dose
Population: All participants who received at least 1 dose of study drug or placebo with evaluable PGEM data at specific time points.
Measure: Mean (Standard Deviation); unit: percentage change in PGEM
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207 | Placebo | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 18
percentage change in PGEM
  0 - 2 hr interval: number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 6 | 11 | 17
  0 - 2 hr interval | 14.4 (35.8) | 18.5 (31.4) | 11.0 (40.6) | -26.6 (25.9) | 17.3 (53.5) | 10.7 (32.7) | -19.8 (36.4) | 5.8 (47.3) | -14.6 (40.7)
  2 - 4 hr interval: number analyzed (Participants) | 8 | 6 | 7 | 7 | 4 | 6 | 7 | 10 | 18
  2 - 4 hr interval | 14.5 (39.4) | -2.1 (43.4) | 5.8 (45.5) | -45.2 (32.3) | 6.1 (66.3) | 29.6 (64.1) | -12.0 (41.4) | 11.2 (32.1) | -30.7 (36.1)
  4 - 6 hr interval: number analyzed (Participants) | 7 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 18
  4 - 6 hr interval | -0.8 (39.3) | -1.5 (57.4) | -22.1 (35.5) | -44.2 (27.3) | -9.2 (56.9) | 15.8 (50.8) | -24.2 (39.4) | 6.3 (44.4) | -32.3 (42.4)
  6 - 12 hr interval | 4.9 (40.9) | -17.9 (56.4) | -13.5 (42.5) | -41.9 (23.7) | -18.8 (42.5) | -13.0 (38.0) | -37.5 (26.2) | 2.9 (44.0) | -36.8 (27.9)
  12 - 24 hr interval: number analyzed (Participants) | 8 | 6 | 7 | 7 | 6 | 6 | 8 | 11 | 18
  12 - 24 hr interval | 3.9 (20.1) | -32.6 (33.5) | -12.9 (31.0) | -37.9 (29.3) | -26.9 (43.6) | -7.3 (38.2) | -43.6 (33.1) | 0.9 (32.8) | -46.5 (17.8)

6. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Urinary Excretion of Prostacyclin Metabolite (PGIM)
Description: The participant's urine was collected during protocol-defined intervals and the PGE metabolite PGIM was assessed. PGIM results for each interval were then compared to the baseline value.
Time Frame: 0 to 2, 2 to 4, 4 to 6, and 6 to 12 hours post dose
Population: All participants who received at least 1 dose of study drug or placebo with evaluable PGIM data at specific time points
Measure: Mean (Standard Deviation); unit: percentage change in PGIM
Groups:
- 450 mg LY3031207 Fed: 450 of LY3031207 administered orally as capsules as a single dose.
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207 | Placebo | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 18
percentage change in PGIM
  At 0 - 2 hr interval: number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 6 | 11 | 17
  At 0 - 2 hr interval | 14.1 (36.5) | 25.2 (41.9) | -3.9 (27.4) | 11.7 (28.0) | 44.6 (44.3) | 137.2 (195.5) | 37.2 (30.1) | -17.0 (24.2) | -18.9 (25.6)
  At 2 - 4 hr interval: number analyzed (Participants) | 8 | 6 | 7 | 7 | 4 | 6 | 7 | 10 | 16
  At 2 - 4 hr interval | 34.0 (64.3) | 30.5 (20.8) | 21.2 (35.4) | 33.1 (42.8) | 244.7 (147.6) | 174.1 (249.0) | 122.5 (114.3) | 6.2 (81.9) | -44.6 (21.3)
  At 4 - 6 hr interval: number analyzed (Participants) | 7 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 16
  At 4 - 6 hr interval | 73.8 (66.1) | 19.3 (45.8) | 31.0 (52.0) | 72.1 (69.3) | 198.3 (80.0) | 186.7 (70.1) | 264.0 (114.3) | 28.3 (71.1) | -25.6 (45.4)
  At 6 - 12 hr interval | 48.0 (45.1) | 52.1 (45.2) | 63.6 (19.1) | 71.7 (66.4) | 208.5 (78.8) | 190.0 (117.5) | 201.4 (141.9) | 57.5 (208.1) | -12.1 (53.8)

7. Secondary Outcome: Pharmacodynamics: Percent Change From Baseline of Urinary Excretion of Thromboxane A Metabolite (TXAM)
Description: The participant's urine was collected during protocol-defined intervals and the PGE metabolite TXAM was assessed. TXAM results for each interval were then compared to the baseline value.
Time Frame: 0 to 2, 2 to 4, 4 to 6, and 6 to 12 hours post dose
Population: All participants who received at least 1 dose of study drug or placebo with evaluable TXAM data at specific time points.
Measure: Mean (Standard Deviation); unit: percentage change in TXAM
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207 | Placebo | 400 mg Celecoxib
Number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 18
percentage change in TXAM
  At 0 - 2 hr interval: number analyzed (Participants) | 8 | 6 | 8 | 7 | 6 | 6 | 6 | 11 | 17
  At 0 - 2 hr interval | -9.0 (10.2) | -5.7 (9.6) | 0.9 (17.4) | -11.3 (10.8) | 4.4 (13.8) | 25.2 (31.5) | 11.0 (24.7) | -11.5 (22.6) | -6.2 (19.3)
  At 2 - 4 hr interval: number analyzed (Participants) | 8 | 6 | 7 | 7 | 4 | 6 | 7 | 10 | 17
  At 2 - 4 hr interval | 4.1 (16.1) | -15.5 (7.7) | 19.7 (23.7) | 0.7 (22.1) | 40.4 (52.4) | 28.3 (58.3) | 106.2 (107.1) | -17.4 (17.2) | -25.4 (17.0)
  At 4 - 6 hr interval: number analyzed (Participants) | 7 | 6 | 8 | 7 | 6 | 6 | 8 | 11 | 17
  At 4 - 6 hr interval | 1.3 (25.4) | -16.5 (11.4) | 1.2 (16.9) | -3.8 (16.4) | 29.4 (29.6) | 16.7 (25.2) | 88.5 (47.9) | -18.3 (18.7) | -33.3 (10.6)
  At 6 - 12 hr interval | 6.8 (29.5) | -15.7 (19.6) | 20.7 (23.2) | 8.0 (25.2) | 30.9 (29.6) | 9.0 (23.1) | 85.8 (85.9) | 13.1 (14.8) | -19.8 (18.3)

ADVERSE EVENTS:
Time Frame: Up To 4 Months
Groups:
- 450 mg LY3031207 Fasted: 450 mg LY3031207 administered orally as capsules as a single dose to participants who were fasted before receiving drug.
Arm/Group | 5 mg LY3031207 | 25 mg LY3031207 | 75 mg LY3031207 | 225 mg LY3031207 | 450 mg LY3031207 Fed | 450 mg LY3031207 Fasted | 900 mg LY3031207 | Placebo | 400 mg Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/8 | 0/7 | 0/6 | 0/6 | 0/8 | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 3/8 | 3/6 | 1/8 | 1/7 | 0/6 | 2/6 | 2/8 | 2/10 | 1/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg LY3031207 (N=8) | 25 mg LY3031207 (N=6) | 75 mg LY3031207 (N=8) | 225 mg LY3031207 (N=7) | 450 mg LY3031207 Fed (N=6) | 450 mg LY3031207 Fasted (N=6) | 900 mg LY3031207 (N=8) | Placebo (N=10) | 400 mg Celecoxib (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gingival infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days